Research Staff Form CMCVAMC IRB
Corporal Michael J. Crescenz VA Medical Center Institutional Review Board

APPROVED by CMCVAMC IRB 2
Date: / 4 / 3 - // 5

TITLE OF RESEARCH PROTOCOL: Reducing Colorectal Cancer Death through Mailed Outreach DATE: 12/16/2015 MIRB# (if applicable) PI Name PI Name Staff Member Name Staff Member Name Staff Member Name Emily C. Paulson, MD, Co-I: Chyke Doubeni, Shivan Mehta, MD, MBA. Adina Lieberman, MPH Kara Magane, MS Name MSCE MD, MPH **MSHP** Emily.Paulson@va.gov Chyke.Doubeni@ Shivan.mehta@ Adina.lieberman@ Kara.Magane@ E-Mail Address uphs.upenn.edu uphs.upenn.edu uphs.upenn.edu uphs.upenn.edu 215-823-5800 x6637 215-823-6333 215-823-6333 215-823-6333 215-823-6333 VA Phone Number 215.662.3349 215-898-9807 Non-VA Phone Number Oversee the development, Oversee the development, Assist with implementing Research Project Manager Research Assistant -Role and Responsibilities implementation, and implementation and and evaluating data -implement study protocol implement study protocol evaluation of the study evaluation of the study 15% 5% 5% 10% 50% % Effort on Study Is this staff member a VA **YES** ☐ YES X YES YES NO T YES □ NO □ WOC ☐ NO employee? □ NO □ NO ⊠ woc ⊠ woc □ woc ⊠ woc Does this staff member YES 
 NO
 NO
 NO exercise independent ✓ YES ☐ YES ☐ YES clinical decision making □NO □ NO ⊠ NO ⊠ NO related to the grant/project? Does this staff member X YES ⊠ YES □ NO come to the CMCVAMC **YES**  YES 
 NO
 NO □ NO and see either VA patients □NO □NO or VA patients' private health information? Does this staff member ⊠ YES decide if potential subjects  $\boxtimes$  YES ☐ YES ⊠ NO ☐ YES ⊠ NO □ NO □NO NO meet inclusion/exclusion criteria? Does this staff member  $\boxtimes$  YES ⊠ YES □ NO obtain subjects' informed X YES ☐ YES □ NO consent? □ NO ⊠ NO ⊠ YES X YES Does this staff member X YES ☐ YES YES

Submit an additional form if necessary.

document in CPRS?

Reminder: All research staff must meet or exceed the minimal standards set forth by CMCVAMC IRB. This form must be updated by the PI and submitted to the IRB for approval before protocol personnel changes can be implemented.

□NO

⊠ NO

⊠ NO

□ NO

R&D Revisions: 07/11/2006; 05/31/2007, 08/14/2008; 03/2009

□NO

| Research Staff Form | CMCVAMC IRB | | APPROVED t | OY CMCVAMC IRB 2 |
|---|---|---|---|---|
| | Corporal Michael J. Crescenz | v VA Medical Center Institutional Review Bo | oard | Date: 12/22/15 |

| TITLE OF RESEARCH P | DATE: 12/16/2015 | | | | |
|---|---|---|---|---|---|
| MIRB# | | | | | |
| (if applicable) | Staff Member Name | Staff Member Name | Staff Member Name | Staff Member Name | Staff Member Name |
| | Kenneth Walton | Danielle Bauscher, MSW | Mounika Kanneganti | Christopher B. Roberts | Amanda Walling |
| Name | | | | | |
| | Kenneth.Walton2@va.gov | Danielle.Bausher@va.gov | mounikak@sas.upenn.edu | Christopher.Roberts5@ | Amanda.walling@va.gov |
| E-Mail Address | | | 1 | va.gov | |
| | 215-823-6333 | 215-823-6333 | 215-823-6333 | 215-823-5800 x 3882 | 215-823-4631 |
| VA Phone Number | | | | | |
| Non-VA Phone Number | | | | | |
| | Research Assistant – | Research Assistant - | Research Assistant - | Dataset Administrator | Program Analyst |
| Role and Responsibilities | implement study protocol | implement study protocol | implement study protocol | | |
| | 15% | 15% | 10% | >1% | >1% |
| % Effort on Study | | | | | |
| Is this staff member a VA | YES | ☐ YES | YES | | ⊠ YES |
| employee? | □NO | □ NO | □NO | □NO | □NO |
| | ⊠ woc | ⊠ woc | ⊠ woc | □woc | □woc |
| Does this staff member | | | | | |
| exercise independent | YES | YES | ☐ YES | YES | YES |
| clinical decision making | ⊠ NO | ⊠ NO | ⊠ NO | ⊠NO | ⊠ NO |
| related to the grant/project? | | | | | |
| Does this staff member | | | | | |
| come to the CMCVAMC | ⊠ YES | ⊠ YES | ⊠ YES | ⊠ YES | ⊠ YES |
| and see either VA patients | □NO | □NO | □NO | □NO | □ NO |
| or VA patients' private | | | | | |
| health information? | | | | | |
| Does this staff member | | | | | |
| decide if potential subjects | YES | ☐ YES | YES | ☐ YES | YES |
| meet inclusion/exclusion | ⊠ NO | ⊠ NO | ⊠NO | NO | ⊠NO |
| criteria? | | | | | |
| Does this staff member | | | | | |
| obtain subjects' informed | ⊠ YES | ⊠ YES | YES | YES | YES |
| consent? | □NO | □NO | NO | ⊠NO | ⊠NO |
| Does this staff member | YES | YES | YES | YES | YES |
| document in CPRS? | ⊠ NO | ⊠ NO | ⊠ NO | ⊠NO | ☐ YES ⊠ NO |

Submit an additional form if necessary.

Reminder: All research staff must meet or exceed the minimal standards set forth by CMCVAMC IRB. This form must be updated by the PI and submitted to the IRB for approval before protocol personnel changes can be implemented.

R&D Revisions: 07/11/2006; 05/31/2007, 08/14/2008; 03/2009

Dear Mr./Mrs. [Last name]

The FIT kit is a simple, effective way to screen for colorectal cancer and takes less than 5 minutes. Here is your FIT (Fecal Immunochemical Test) kit for colorectal cancer screening at no cost to you.

### Why is this important?

yourself cancer free By completing the FIT screening every year, you are taking an important step toward keeping

### How do I use the kit?

the kit and remember to write your name, date of birth, and the date you completed the test on the bottle. Mail back the kit within 48 hours in the self-addressed, pre-paid envelope included movement. You only need one sample to complete the screening. Follow the instructions included in Place the kit in your bathroom and collect a stool ("poop") sample the next time you have a bowel

#### What is next?

results, it may be necessary to come in for further testing of your FIT screening, and I will let you know the results as soon as I have them. Depending on your There is no need to call to let me know that you completed the test. The lab will send me the results

### What if I have questions?

phone number and a time to contact you Fridays. If you call and nobody is available to answer the phone, please leave a message with your team at 215-615-4796. Staff are available to help you from 8AM to 5PM on Mondays through If you have any questions before, during, or after completing the FIT, please contact our screening

I hope you complete this free and important screening test.

Sincerely,

[[Doctor's Name]] [[Title]]

**CMC VA Medical Center** 



[[Patient first name]] [[last name]]
[[street address]]
[[city]], [[state]] [[ZIP code]]

[[date]]

Dear Mr./Ms.[LASTNAME]:



You will get your screening kit in an envelope within 1 to 2 weeks.

privacy of your own home. convenience, we will mail you a FIT kit at no cost to you. FIT stands for Fecal The kit has everything you need to complete your part of the screening in the Immunochemical Test - a simple, effective way to screen for colorectal cancer. Our records show that you are due for colorectal cancer screening. For your

# Colorectal cancer is very curable when found early.

cancer free. Depending on your FIT results, I may need you to come in for further By taking this test every year, you take an important step toward keeping yourself

# Completing the FIT takes less than 5 minutes.

Full instructions are provided in the kit. need only one stool ("poop") sample, and do not need to do anything to prepare The FIT kit will be in your mailbox within 2 weeks at no cost to you. You will You will mail the kit back to the VA using a self-addressed, pre-paid envelope.

# Colorectal cancer can run in families.

If this is the case for you, let's talk about the best way for you to be tested and how

another reason that you no longer need screening, please call our screening team at 215-615-4796 and we will update your records. If you get your colorectal cancer screening tests outside of the VA, or if there is

Sincerely,

[[Doctor's Name]][[Title]]
CMC VA Medical Center



```
[[Patient first name]] [[last name]]
[[street address]]
[[city]], [[state]] [[ZIP code]]
```

## Dear Mr./Ms.[LASTNAME]:

you should get screened for colorectal cancer. our screening team at 215-615-4796 to schedule an appointment to discuss how Our records show that you are due for colorectal cancer screening. Please contact

# Colorectal cancer is very curable when found early.

to come in for further testing. free. Depending on the test you receive and the result of that test, I may need you By getting screened, you take an important step toward keeping yourself cancer

# Colorectal cancer can run in families.

If this is the case for you, let's talk about the best way for you to be tested and how

and we will update your records. reason that you no longer need screening, please call our office at 215-615-4796 If you get your colorectal cancer tests outside of the VA, or if there is another

Sincerely,

[[Doctor's Name]][[Title]]
CMC VA Medical Center



#### Please fill out the following information so that we can ensure we have the most accurate information in your medical record at the VA.

Below are types of screening for colorectal cancer. For the test(s) that you

| have received, please check | the box and write the date you had the test(s) |
|---|---|
| ☐ I have not received any | colorectal cancer screening tests |
| ☐ Stool test <sup>1</sup> | Date: |
| ☐ Colonoscopy <sup>2</sup> | Date: |
| ☐ Sigmoidoscopy <sup>3</sup> | Date: |
| ☐ CT Colonography <sup>4</sup> | Date: |
| If you have any questions, | please call us at 215-615-4796. Thank you! |
| Name (print): | Date: |

- Stool test, called either FOBT (Fecal Occult Blood Test) or FIT (Fecal Immunochemical Test) are tests where the patient collects 1 to 3 stool or "poop" samples at home and sends them to a lab to be tested for hidden blood.
- Colonoscopy is a procedure that lets a doctor closely look at the inside of your bowels for signs of colon cancer by inserting a small tube into the rectum. Patients are usually given medicine to help them relax and sleep while it's done.
- Sigmoidoscopy is a procedure that allows a doctor to look closely at only the lower part of the colon and the rectum. To do this, the doctor inserts a thin (about the thickness of a finger), flexible, hollow, lighted tube into the rectum. The patient usually doesn't need medicine to help them relax.
- CT Colonography is a special x-ray of the large intestine, which includes the colon and rectum. To do this, the doctor inserts a well-lubricated tube into the rectum. The patient usually doesn't need medicine to help them relax.

APPROVED by CMCVAMC IRB 2
Date: 12/37/15

### Content Requirements for IRB Committee CMCVAMC Specific Protocol Summary

### **CMCVAMC IRB**

Corporal Michael J. Crescenz VA Medical Center Institutional Review Board

- Protocol Title
- Full Protocol Title: heuron's Screening
  Screening
  Date of Protocol Summary and Version #: Version 7 December 16, 2015
- œ Principal Investigator's Full Name and Degree: E. Carter Paulson, MD, MSCE
- ? Co-Investigator's Full Name and Degree: Chyke A. Doubeni, MD, MPH; Shivan Mehta, MD, MBA
- D. Pennsylvania to support pilot data collection on this project. Merit on the next funding round. We currently have funds from CHERP and the University of feasibility of the screening program, and doing so will enable us to apply for a full HSR&D conduct the study, even if a favorable funding decision is not received, to assess the requirements. An IRB protocol under review is a condition of funding. However, we wish to SMRB. HSR&D intends to fund this proposal upon successful completion of all Just-in-Time Financial Sponsor: This proposal was reviewed at the August 2015 meeting of the HSR&D
- Ш Grant: N/A
- П Protocol Number: PPO 14-369
- G
- Institution(s) responsible for the project:

  1. For single-site studies CMCVAMC is the only institution involved. Yes ⊠ No □
- For multi-center studies.
- No N/A CMCVAMC is the Coordinating Center in which the PI is the lead investigator. Yes
- Provide the name of the Coordinating Center. Yes ☐ No ☐ N/A ☐
- List the name of the other sites involved.
- Provide the FWA numbers for each of the other sites involved

## THE FOLLOWING INFORMATION MUST BE CMCVAMC-SPECIFIC, WHAT WILL BE DONE WITH CMCVAMC-RECRUITED VETERANS. THAT IS, SPECIFIC TO

as well as barriers to screening uptake among veterans is not well unknown, and there are potential disparities that remain undiscovered. The U.S. Preventive Services Task Force, as adults to 80% by the year 2018. Reports suggest that the VA has already achieved this screening target. However, much of the existing knowledge on CRC screening in the VA has been on veterans who have had recent VA healthcare visits. Thus, the true rate of screening Background and Significance: Colorectal Cancer (CRC) is the second leading cause of does the Veterans Health Administration (VHA) Directive 2007-004, recommends screening Cancer Roundtable launched an initiative to increase CRC screening uptake among eligible mortality rates for CRC over the past three decades. Recently, the National Colorectal increasing uptake of screening has been a key contributor to the declining US incidence and 100,000 persons by 2020. Screening is cost-effective for preventing CRC death. The VA, which dovetails into the US national objective to reduce CRC mortality to 14.5 per cancer deaths in the United States (US). CRC prevention and control is thus a priority for the

by improving the screening process. Thus, the proposed project is specifically geared access to and use of effective screening among all veterans, particular those hard to reach, screening by direct mailed outreach. towards simplying the screening process by changing the default approach to initiating health care visit and a provider's recommendation. This application seeks to create a pilot program of population-based mailed FIT outreach for CRC screening in the VA with the levels such as the need for a face-to-face encounter. The long-term goal is to optimize potential for widespread adoption to overcome barriers at patient, provider and systems disparities. Two of the strongest predictors for receiving CRC screening are having a regular populations such as racial minorities, even in the VA, contributing to incidence and mortality every 10 years as equally acceptable strategies. CRC screening is underutilized in some sigmoidoscopy every five years with mid-interval gFOBT or FIT, or optical colonoscopy occult blood tests (gFOBT) such as the fecal immunochemical test [FIT) annually, flexible for CRC in average-risk 50-75-year-old adults using highly sensitive guaiac-based fecal

data linkages to, in future studies, enable evaluation of FIT performance characteristics and screening to eligible veterans through multilevel interventions. We will also create electronic specifically address the need to identify and remediate potential failures to identify and offer not rely on having a clinical office visit. As shown in the conceptual framework (Figure 1), we implementing and disseminating a pilot mailed-FIT screening outreach program that does study and improve the delivery and effectiveness of CRC screening in the VA by developing, help close critical evidence gaps for optimizing screening among veterans Purpose of the Project: This application seeks to establish the foundation to systematically

Figure 1: Conceptual framework for optimizing the VA screening process for this pilot project



- <u>ب</u> having an office visit, by conducting a proof-of-concept 3-arm parallel-design pragmatic in the Corporal Michael J Crescenz VA Medical Center (CMCVAMC) that does not rely on development, implementation and dissemination of a mailed FIT outreach program in the CMCVAMC that does not rely on having an office visit. The main study aim is to develop, assess feasibility of a population-based screening outreach approach through the Describe the Research Questions or Hypotheses: As this is a pilot study, the focus is to randomized trial to: implement and disseminate a pilot population-based mailed FIT outreach screening program
- Compare the effects of usual care (UC), screening invitation + reminder (invitationreminder), or screening invitation + mailed FIT kit + reminder (mailed-FIT)
- Explore whether the FIT completion rate varies by age or race/ethnicity


- Explore barriers to use of mailed outreach screening for veterans
- <u>.</u> ~ Primary Outcome Variable(s): The primary outcome is the completion rate of FIT within 6 months of baseline.
- ŗ screening test within 6 months of baseline Secondary Outcome Variable(s): Our secondary outcome is the receipt of any CRC

| | | | | | <u>.</u> |
|---|---|---|---|---|---|
| 'n | | | | | ş |
| De | Ò. | | <u>a</u> | S | φ |
| Design: | If yes, this study must be registered on Cli | NOT APPLICABLE (Pilot) | <ol> <li>If yes, what type? Check all that apply.</li> </ol> | 1. Is this a clinical trial? ☐YES ⊠NO | M. Study Design and Methods: |

What research methods will be used in the project? Check all that apply.

| Other (Describe) | Specimen Collection | ☐ Control Group | Focus Groups | Behavioral Observations | |
|---|---|---|---|---|---|
| | Deception | ☐ Placebo | □ Randomization | Chart Reviews | |
| | ☐ Telephone Survey | Withhold/Delay Treatment | ☐ Double-Blind | ☐ Video Taping | ☐ Audio Taping |

- ġ. effect of usual care (UC), and population-based screening invitation + reminder (invitation-reminder only), or screening invitation + mailed FIT kit + reminder (mailedconduct a 3-arm parallel-design pragmatic randomized trial to compare amongst the three arms. FIT). The 3,388 potentially eligible veterans will be block-randomized to one of the Describe how randomization or other treatment assignment will be made: We will
- ဂ prior to selection, are due for CRC screening, and are asymptomatic for the study but who, have not been seen by primary care in the past 18 months years old, have received care in CMCVAMC in the 18-48 months prior to selection Pennsylvania and Southern New Jersey who, during the funding year, are 50 to 75 via CPRS chart review; eligible veterans include veterans in the southeastern 1, 1999 through December 31, 2008): We will identify all potentially eligible veterans For retrospective research studies, provide the "look-back" period. (e.g., December

### Study Duration:

- October 1, 2015 (or as soon as Approved by the IRB) to September 30, 2016. Provide the estimated length of time to enroll all subjects and complete the study.
- Ö study will primarily test the effect of an outreach mailing, along with reminders, of the mailing the kits through Months 3-5 and will conclude follow-up procedures by Month FIT to veterans. The outcome will be assessed through Months 3-7. We anticipate Explain the expected duration of subject participation including any follow-up: This 11 of the study period.
- ဂ of completion is December 31, 2016. Specify the projected date of completion of the proposed study. The projected date
- Drug Information: NOT APPLICABLE
- Specify if the drug or biological agent is:
- FDA approved:
- Used for off-label purposes
- iii. Not yet FDA approved.

- 6 and off-label drugs, biological agents or nutritional supplements: Include the FDA Investigational New Drug (IND) number for all non-FDA approved
- 0,0 Provide all relevant information about the drug
- medications not permitted while enrolled in the study. Explain any wash-out periods, rescue medications permitted and any type of
- θ Describe blinding and un-blinding procedures.
- information on any drug used for research purposes. Include the dosage, route of administration, previous use, and the safety and efficacy
- ġ. Describe rationale for the dosage in this study.
- ħ knowledge. Justify why the risks are reasonable in relation to anticipated benefits and/o
- Describe where drug preparation will be done. All drugs for CMCVAMC subjects must be dispensed through the VA investigational
- Describe where the study treatment will be administered.
- Describe plan for tracking a non-compliant treatment study subject
- 3 Summarize any pre-clinical data.
- investigational drug. Describe the process for the storage, security, dispensing and return of an

### 5 Investigational Device: NOT APPLICABLE

- ä significant risk devices and if an IDE exists for a non-significant device. The Investigational Device Exemption (IDE) number must be submitted for all
- 6 specify whether or not the sponsor has determined this device to be a "significant Significant Risk or Non-significant Risk - If a device is not approved by the FDA, risk" or "non-significant risk" as defined by the FDA.
- 0.0 Provide all relevant information about the device.
- Describe blinding and un-blinding procedures
- e. Specify if device is:
- FDA approved
- Used for off-label purposes
- Not yet FDA approved.
- Investigator or Pharmacy Services. Explain if the investigational device will be delivered and/or stored by the Principal
- g. investigational device. Describe the process for the storage, security, dispensing and return of an
- ħ. For research involving an investigational device, describe the SOP or plan for device
- :associated with the protocol will have access to the device. Address how the device will be stored in such a way that only research staff
- ÷. used in participants of this research protocol. Describe measures that will be put into place to ensure that the device will only be

| Does |
|-------------------------------------|
| this |
| s project involve international rea |
| ect ii |
| lovr |
| e<br>F |
| itern |
| ation |
| <u>าล</u> |
| sea |
| rch? |
| j |
| YES |
| $\boxtimes$ |
| $\overline{z}$ |

#### 0 Study Procedure

Study Procedures: We will conduct a 3-arm parallel-design randomized trial to compare sections below (Figure 2). mailed FIT kit (mailed-FIT). The program flow is outlined below and described in the UC, screening invitation + reminder alone (invitation-reminder), and invitation-reminder +

HRPP Approval: <u>06/15/2011</u>
R&D Approval: <u>07/05/2011</u>
File: K: New IRB Forms



- of the registry in subsequent calendar years to minimize mailing FIT to veterans who are already up-to-date. Individuals will age into (as they turn 50) or age out of (age >75) the earlier ages (i.e., ≥45 years) to expedite outreach as they approach the eligible age. registry. In the future, we will explore the possibility of adding veterans to the registry at the beginning of 2016. We will develop an approach to update and improve the accuracy months prior to the start of our study and not currently up-to-date on CRC screening in identify age-eligible veterans who had received medical care at CMCVAMC in the 18-48 the CMCVAMC. At the start of the pilot program, we will run the electronic query to We will build on the database currently used by Dr. Dubb (consultant) to monitor FIT at Creation of Tracking database: A database of eligible veterans is critical to the program.
- ω Society. We are currently working on procedures to pre-label kits with each participant's instructions in English and Spanish using resources developed by the American Cancer about 1 week after the screening invitation. The kit will have specimen collection adapt their outreach materials – see attached for examples). The FIT kit will be sent practiced in Kaiser Permanente Northern California (we have received permission to signed pre-notification letter and a screening confirmation card will precede the kits, as unique information. Mailing the FIT kits: In the mailed-FIT arm, a screening invitation that includes a PCP-
- 4 will be conducted at 6 months from baseline on all participants to ask for information on history in VistA with both EMR and patient interview. The screening history questionnaire screening use. We will conduct formal chart review on the study sample (n=783). At the and administrative data may underestimate, and patient report may overestimate, the test was performed – interviews at baseline will contaminate the UC arm. We have receipt of CRC screening test, the last test and type (if applicable), and location where end of the study, we will also conduct surveys of participants to compare their screening we will test the accuracy of electronically determined screening histories. Chart audits incomplete, because tests received outside the VA may not be recorded in VistA. Thus, identify CRC screening history in EMR. The advantage in the VA is its integrated delivery structure. However, the screening history in CPRS (a Veterans Health Information Systems and Technology Architecture [VistA] computer application) may be Validation study of screening history. We have extensive experience in algorithms to

- accuracy of algorithms to determine guideline-concordant screening by identifying among 783 subjects). This will allow us to refine our program strategy and improve 80% power to detect 3.8% false negative rates (that is, if 30 were previously screened have extensive tools of our own to use for chart audit and patient surveys patient and registry level predictors that are correlated with false negative rates. We
- Ġ of this approach. evaluation. We will, in future studies, develop procedures to evaluate the effectiveness risk factors. Doing this will allow the latter group to be directed to their doctor for information cards in the invitation letters about CRC symptoms, family history, or other Distinguishing asymptomatic participants from those with GI symptoms: We will provide
- 9 procedures. We will safeguard participant data during and after mailing. Specimen analysis: The OC-FIT CHEK is analyzed at the CMCVAMC using OC Sensor assure that we can contact screen-positive participants, we will obtain updated contact approaches such as returned receipt confirmation. To support annual rescreening and information such as telephone numbers and emergency contacts, as part of the outreach veterans. We will assess the extent to which kits are successfully delivered and explore Valid contact information is critical to the program, but may be challenging with some
- 7. ≥100ng/dL. The machine records (but does not report) the quantitative results of the hemoglobin. Results are provided as positive if the hemoglobin concentration is for future studies. hemoglobin concentration in the sample, which we will seek to obtain from the laboratory according to manufacturer's instructions to minimize potential degradation of concentration of hemoglobin in the collected sample. Specimens will be analyzed DIANA, an auto-analyzer system that provides quantitative results corresponding to the
- Ω Patients who test positive will be notified by mail and phone. We will track results with positive results by phone, as needed, and by monthly CPRS queries and EMR review until diagnostic testing is completed or clinical decision is made not to do diagnostic using existing procedures. Patients with a negative result will be informed by mail. recorded in CPRS and the tracking REDCap database and communicated to the PCP Communication of results and diagnostic work-up for abnormal screen: Results will be
- 9 to ambient temperature exposures. ongoing studies, to enable us to monitor performance characteristics variation according Oceanic and Atmospheric Administration (NOAA) public databases, as we have done in date as the standard. We will also develop an approach to create linkages to National positive of FIT for detection of CRC using detection of CRC within 24 months of result and tumor stage, morphology, histologic behavior characteristics, grade, and location (subsite) using International Disease Classification, Oncology codes. Potential analysis approximately 120 VAMCs. Our VACCR application will request CRC diagnosis dates, for this exploratory study will examine the sensitivity, specificity, and the predictive value patient-level and environmental factors. The VACCR aggregates data collected by detection of CRC at the VA, including FIT's performance variations according to selected study patients to enable full evaluation of performance characteristics of FIT for the Data Linkages: We will apply for VA Central Cancer Registry (VACCR) linkages on all
- Study Procedures for the Proof-of-Concept Pragmatic Trial: We will conduct a 3-arm from ongoing practices at the CVMAC and separately from standardized invitation and determine if mailed invitation with a FIT kit is effective at increasing uptake separately screening invitation + mailed FIT kit + reminder (mailed-FIT). The rationale is to parallel-design pragmatic randomized trial to compare amongst the effect of usual care (UC), and population-based screening invitation + reminder (invitation-reminder only), or


- veterans screening behaviors. reminders. Ongoing evaluation of these approaches will help VA adapt to changes in
- 11. Recruitment. An estimated 783 eligible patients will be recruited for this trial. We will obtained a waiver of informed consent from the IRB since this is considered minimal risk criteria. There are an estimated 3,388 potentially eligible veterans for this pilot. We have support from Dr. Tzanis, for participation and to confirm the inclusion and exclusion obtain PCP approval, through discussion at schedule clinical and program meetings with to the participants, and obtaining consent would inherently change the intervention.
- 12. Randomization: Patients will be block-randomized to UC, invitation-reminder, or mailedprior to mailing invitations to study participants.

  a. Participants randomized to UC: These patients will continue to receive the current all study materials to patients during Months 3-5 of the study in weekly waves of about 50 mailings; with this volume, it is feasible for us to confirm eligibility through chart audits FIT with guidance from Dr. Richardson to achieve the desired sample size. We will mail
- participants in the trial, including those in UC, will receive follow-up of test results and will be embedded within this existing program for a pragmatic approach. However, all practice at CMCVAMC of offering screening during an office visit. Other interventions navigation to diagnostic colonoscopy for positive FIT results.
- b. when participants cannot be reached by phone and track the success of each veteran may be homeless. Thus, we will also explore sending mailed reminders approach used during the study. change or run out of purchased minutes, but addresses may also change or a effective at reaching veterans than phone calls because telephone numbers may was sent (time zero). It is generally unclear whether mail reminders may be more For the purposes of this intervention, Week 1 will be the week the invitation letter will also receive notification of test results and navigation to colonoscopy, if needed. receive three weekly reminders at weeks 4, 5, and 6 from the invitation letter. They screening is not completed (even if they have an appointment scheduled). They will inform patients that a telephone reminder will follow in 4 weeks from invitation letter if he/she is not eligible and to update the contact information on record. The letter will confirmation card and instructions to contact the study team if the patient believes as change in bowel habit with rectal bleeding. The packet will also have a screening offered at CMCVAMC), and symptoms that should prompt diagnostic work-up such such as FIT and colonoscopy and, if appropriate, Cologuard (sigmoidoscopy is not see below). The information will include lay-audience description of screening tests Participants randomized to screening invitation-reminder: These patients will information about CRC testing in the mail-FIT arm (except the kit and instructions, continue to receive UC. They will in addition receive an invitation letter with all of the
- 9 additional calls at the end of weeks 5 and 6, if needed.82 For the purposes of this an appointment scheduled, as with the invitation-reminder arm), followed by 2 notification letter was mailed will receive a live telephone reminder (even if they have completed. Patients who do not return their kit after 4 weeks of the date the preand instructions to contact the study team if the patient believes he/she is not eligible and to update the contact information on record. They will be informed that a We will explore and evaluate the approaches for successfully contacting participants intervention, Week 1 will be the week the pre-notification letter was sent (time zero). telephone reminder will follow 4 weeks from notification letter if screening is not week later (see section D2d2). Patients will receive a screening confirmation card Participants randomized to Mailed-FIT will receive a mailed FIT pre-notification letter in our study setting (plus a screening invitation and screening confirmation card) followed by the kit 1


- selection, are due for CRC screening, and are asymptomatic for CRC. Pennsylvania and Southern New Jersey area who, during the study period, are 50 to 75 years old, have received care in CMCVAMC in the 18-48 months prior to selection for Study Population: The study population will be all veterans in the southeastern the study but who have not been seen by primary care in the past 18 months prior to
- 14. Setting: This study will be conducted at CMCVAMC in southeastern Pennsylvania and Southern New Jersey.
- 15. Exclusion: We will exclude tests of patients with known gastrointestinal symptoms such exclude patients with evidence of prior colonoscopy within 10 years, sigmoidoscopy 3,388 veterans to draw from for our study based on screening eligible population at the within 5 years, and FOBT/FIT in the same calendar year. There is a pool of at least Disease (9th and 10th edition) diagnostic code or by self-report (Figure 2). We will as bleeding, unexplained weight loss, or change in bowel habits, family history of CRC, inflammatory bowel disease (IBD), or colectomy using International Classification of
- CPRS/Regional Data Warehouse Test results: Data on the date, and result of FIT performed will be obtained from
- 17. Measurement of Outcome: The primary outcome measure in all analyses is the an adequate sample size to obtain meaningfully precise estimates. several of those factors to be considered as covariates in some analyses as shown in reminders, positivity rate, completion of diagnostic colonoscopy. We will measure of other outcomes, including the proportion of non-responders who responded to diagnostic testing, we will define a third outcome as receipt of screening plus timely diagnostic testing (within 90 days) when positive. We will also collect data on a number such an alternative definition will include those who received a colonoscopy for any test in the 6-month period after enrollment into the study. Our rationale as articulated in Gupta et al.,39 is that the 'best test is the one that gets done'. Thus, the numerator for Table 1, recognizing that some of these variables will be exploratory, as we will not have indication. Since the screening process for a positive tests is completed only after We will also evaluate a secondary outcome measure of receipt of any CRC screening completion rate of FIT within 6 months of the mailing of the screening invitation. Absence of screening completion data in CPRS will be recorded as failure to complete screening.
- outcome measures. analyze an 'any CRC screening test' outcome, and the other pre-specified secondary outcome data because outcomes will be tracked in integrated electronic medical mailed-FIT and invitation-reminder are equal using an "intention-to-treat" approach, based on a 2-sided alpha of 0.05. We do not anticipate loss to follow up or missing Analysis plan on primary outcome measures to compare the effects of UC, invitationrecord systems. We will examine the distribution of test types to assess the ability to hypothesis that the completion rates between the mailed-FIT and UC and between reminder, and mailed-FIT): We will use Chi-squared statistic to test the null
- Þ VA study found that screening use differed by age and was lower among persons of black race. We will model fit completion by race/ethnicity (African Americans vs. needed. We will use both univariate and multivariable logistic regression analyses (2. to be targeted when a program is fully implemented and if larger sample sizes will be effect modification. This analysis will allow us to understand if specific groups need interaction terms, to explore the overall effect of race/ethnicity and age, and possible others), age (50-64 vs. 65+), and race/ethnicity\*intervention and age\*intervention variable) among all study participants using logistic regression. Our rationale is that a the association of age and of race/ethnicity with the FIT completion rate (dependent Exploratory analysis of FIT completion rate by age or race/ethnicity. We will assess


- additional analyses will be restricted to those with valid addresses. sided alpha of 0.05). The primary approach will be 'intention-to-treat' analysis and
- ဂ dates and CRC diagnosis ascertainment. the FIT positivity rates and explore the relation with CRC diagnosis using 2 X 2 contingency tables as described section D2d8, using 1 or 2 years between FIT result explore the number of cases of CRC diagnosis in CMCVAMC patients and assess by calling non-responders. Once tumor registry linkage is established, we will seek to seek to verify addresses and assess our ability to contact study veterans by phone the proportion of participants whose mail was returned due to bad addresses. We will Exploratory analyses of mailed outreach screening barriers: A valid participant contact information is key to a successful outreach. Thus, we will track and assess
- a ineligible post-randomization, we will identify about 783 patients for this trial. vs. mailed-FIT. Accounting for the possibility that up to 20% of participants could be 152 patients per arm will give a power of 80% for the screening invitation-reminder 500 (250 per arm) will give 80% power for UC vs. screening invitation-reminder, and reminders, and 40% with mailed-FIT. With those assumptions, a total sample size of analysis, we assumed 15% screening rate in UC alone, 25% with invitationcompleted screening compared to 12% in UC.38 In our power and sample size that, among underserved patients in Dallas, 40% of those assigned to mailed-FIT Sample size and power estimates for primary outcome measures: Gupta et al. found
- 18. Explain if and how the follow-up of subjects will occur. All participants, including and phone call from trained staff to explain the findings and assist in scheduling a colonoscopy within 30 days in collaboration with the CMCVAMC gastroenterology 2). Participants who test positive (estimated 4-6%, or 31-47 patients) will receive a letter record the data into the tracking REDCap database with guidance from Dr. Dubb (Figure staff will send the patient a letter with the results (and education about future testing) and funding availability. All returned kits will be analyzed as described in section D2d6. Study electronically over a minimum of 12 months from the invitation date, depending on screening after invitation or pre-notification letter, but our goal is to track outcomes outcomes. We will set a minimum of 6 months from time zero to determine completion of batches each week, so that even those in UC will have a set reference date for tracking those in UC, will be tracked electronically in VistA. We will select randomized patients in
- 19. Describe where, how and who will be conducting study procedures. The study will who are Co-Investigators on this study. Drs. Dubb and Tzanis will serve as consultants. will oversee all research activities in collaboration with Drs. Richardson and Doubeni guide them on scheduling a colonoscopy. In addition, a research assistant will call patients with a positive result to inform and assistance in completing the kit will be contacted to support them in completing the test kits or complete screening in a timely manner. Also, some participants needing trained research assistants will contact patients by phone if they do not return the test All study activities will be logged into secure REDCap databases at the CMCVAMC. The be conducted under the auspices of CHERP using trained research assistants. The PI
- interviews at baseline will contaminate the UC arm. These surveys take 10-20 the last test and type (if applicable), and location where the test was performed baseline on all participants to ask for information on receipt of CRC screening test interview. The screening history questionnaire will be conducted at 6 months from participants to compare their screening history in VistA with both EMR and patient complete the questionnaires/tools. At the end of the study, we will conduct surveys of If a survey study, specify the estimated amount of time that subjects will need to


Ф If a blood draw, specify the amount of blood to be drawn in milliliters and in drawn. Not Applicable teaspoonfuls or tablespoonfuls and specify how often and where the blood will be

# 20. Data Collection (Include all questionnaires and survey tools with the submission)

- screening history questionnaire will be conducted at 6 months from baseline on all interviews: At the end of the study, we will conduct surveys of participants to compare their screening history in VistA with both EMR and patient interview. The instrument is included in the submission. type (if applicable), and location where the test was performed. The survey participants to ask for information on receipt of CRC screening test, the last test and Provide the mode of data collection, e.g. telephone, in-person, questionnaire,
- ō with guidance from the PI and Drs. Richardson and Doubeni. The research data obtained will be stripped of all identifiers prior to analysis at the CHERP. research assistants under the supervision of the PI in collaboration with Dr. Doubeni. The Dataset Manager and/or the Statistical Analyst will perform analysis on the study for a complete outline of how data is collected. Data collection will be performed by Provide the precise plan for how data is to be collected or acquired. See section 12
- ? Primary Care Clinic. Data entry will take place at: Exact location where data will be collected: Data will collected at the CMCVAMC

Center for Health Equity Research & Promotion

3900 Woodland Avenue, Room 236, Cubicle #9 Philadelphia VA Medical Center Annex

Philadelphia PA 19104

- <u>a</u> investigator, research coordinator. The "title" of individual(s) collecting the data and analyzing the data, e.g. principal
- E. Carter Paulson, MD, MSCE, Principal Investigator Chyke A. Doubeni, MD, MPH, Co-Investigator
- Shivan Mehta, MD, MBA, Co-Investigator
- <u>.</u> Christopher Roberts, MPH, Data Set Manager
- Statistical Analyst (TBD)
- Φ. Provide a time line for each aspect of the study. The timeline is shown in the Figure

Dissemination of results Conduct analysis on study aims Apply for additional funding Exploratory: initiate VACCR linkages Evaluate response rates to mailed FIT outreach Send screening reminders to participants Mail FIT outreach kits to participants 1a. Send screening invitations to participants Design the program AIM/Objective Evaluate barriers of using mailed outreach screening for veterans Test algorithms Months
1 2 3 4 5 6 7 8 9 10 11 12

Figure 3: Timeline and milestones

# 21. Chart/Records/Data Review (retrospective and/or prospective):

- Provide the planned or approximate number of charts/records/data to be accessed
- CMCVAMC: 783
- Other site: NOT APPLICABLE
- ġ. Does this protocol employ an Honest Broker? ☐YES ⊠NO
- If yes, provide name of individual


- Research Assistants will access the charts. If no, explain who will access the charts/records. The PI, co-Investigators and the
- Describe from what database charts/records/data will be accessed. Charts will be accessed through CMCVAMC CPRS/VistA

# 22. Future Use of Data and Re-Contact, if applicable.

- research, the following information must be provided to the participant:

  i. Where will the data be stored? The data will be stored in the CMCVAMC clinical If any of the participant's data are going to be retained after the study for future
- dual microprocessors (for a total of eight processors) and 32 gigabytes of RAM. a redundant array of independent disks. This virtual server resides on a 64-bit Dell PowerEdge physical machine running four Intel Xeon X5460 3.15GHz 64-bit Information Security Management Act (FISMA) standards. The servers reside behind the VA firewall and are entirely compliant with Federal server running 30 gigabytes of RAM, and 2.2 terabytes of disk space located on (CHERP's) secure analytic servers. CHERP has a 64-bit Windows 7 virtual performed/stored on Center for Health Equity Research and Promotion's All analytic data will be stripped of identifiers. All data analyses will be REDCap databases. Analytic Datasets will be stored in VA databases at CHERP
- Manager/Analyst, and Research Assistants Who will have access to the data? The PI, Co-Investigators, Statistician, Dataset
- Ö. informed consent document must contain this information. Not applicable. Results medical care will be provided to patients during the course of the study as happens in routine screen. If subjects will receive aggregate study results at the end of the study, the re-contact patients in future studies to assess the response to annual invitation to participant would be re-contacted whether within the VA or outside the VA. We will If the subject is going to be re-contacted in the future about participating in future research, this must be specified. Describe the circumstances under which the

### 23. Specimen Collection:

- a. based colorectal cancer testing. This is collected for diagnosis of colorectal cancer. treatment or diagnosis: Stool sample (from a bowel movement) is collected for stool-Give the source of all specimens and whether they were collected for research
- Ö. the specimens will be at the discretion of the CMCVAMC laboratory; Room 3b123 State where specimens will be stored, secured and when discarded. Disposition of
- S the specimen collection is part of routine care Explain how destruction of samples will be substantiated. Not applicable because

### P. Genetic Testing:

- has predictive value. Not Applicable specific disease or condition, but at this point it is not clear if the genetic marker Explain if the study is looking for an association between a genetic marker and a
- studies in this category will not involve participant counseling. The uncertainty regarding the predictive value of the genetic marker is such that
- ġ. predicting the development of that specific disease or condition. and a specific disease or condition is such that the marker is clinically useful in Describe if the study is based on the premise that a link between a genetic marker

| | ဂ |
|---|---|
| ☐ Yes [ | Will the |
| | subject t |
| □<br>N<br>A | be notified |
| | of the re |
| | esults a |
| | nd the p |
| | provision |
| ( | for g |
| | enetic |
| ( | c. Will the subject be notified of the results and the provision for genetic counseling? |

- d. If yes, explain further.
- If biological specimens are used in this protocol, please respond to the following questions by checking the appropriate box:


| <b>!</b> | .∸ <u>B</u> | | |
|---|---|---|---|
| Property of the control of the contr | c. b. a. | 9 | |
| <ol> <li>Provide the planned or targeted enrollment at: <ul> <li>a. CMCVAMC - 783</li> <li>b. Other sites - Not applicable</li> <li>c. Not applicable; chart review or use of previously collected data</li> </ul> </li> <li>Screening and/or Eligibility Requirements <ul> <li>a. Describe and provide justification for.</li> </ul> </li> </ol> | <ol> <li>Banking of Collected Specimens: <ol> <li>Will collected specimens be banked? □YES □NO □N/A</li> <li>IF BANKING SPECIMENS, IT MUST BE AT AN APPROVED VA REPOSITORY. (For additional information, refer to VHA Handbook 1200.12, Use of Data and Data Repositories in VHA Research - March 9, 2009.)</li> <li>If yes, specify the location where specimens will be banked.</li> <li>If the location is a non-VA site, has the mandatory approval from the Chief Officer of Research and Development (CRADO) been obtained through submission of a tissue banking application (VA Form 10-0436 - Off-site Application for an Off-site Tissue Banking Waiver)? □YES □NO □N/A</li> <li>If applicable, attach a copy of the VA Form 10-0436</li> <li>Explain how destruction of banked samples will be substantiated.</li> </ol> </li> </ol> | Will specimens be de-identified? ☐YES ☐NO ☐N/A i. If yes, please describe the procedures to be used. ii. Include at what point in the process the specimens will be de-identified. Describe what measures will be taken to minimize the following risks from breaches of confidentiality and privacy resulting from participating in This aspect of the research project: i. physical ii. psychological iii. financial iv. social v. legal harm | Does the project involve genetic testing? Will specimens be kept for future, unspecified use? Will samples be made anonymous to maintain confidentiality? (Instructions: Note: If there is a link, it is not anonymous. Coding is not anonymous. Will specimens be destroyed after the project-specific use is completed? Will specimens be sold in the future? Will subjects be paid for their specimens now or in the future? Will subjects be informed of the results of the specimen testing? Are there any implications for family members based on specimen testing results? (If yes, they may be participants.) Will subjects be informed of results obtained from their DNA? |
| | IEPOS<br>If Data<br>In the (<br>In subn | lentifiers from the sect of th | |
| | and L<br>Chief (<br>nission<br>an Ot | n brea<br>the | |
| | <i>∑Ata</i> Dafficer Officer of a ff-site | iches | |

Q


Ά,

- the CMCVAMC includes the period during which 3-sample testing was being regularly used at prior to selection, are due for screening, and are asymptomatic for CRC. This for the study but who have not been seen by primary care in the past 18 months 75 years old, have received care in CMC in the 18-48 months prior to selection Pennsylvania and Southern New Jersey who, during the funding year, are 50 to Inclusion criteria: The pragmatic trial will include veterans in southeastern
- <u>=</u>: information used to exclude patients will be derived from the electronic queries or sigmoidoscopy within 5 years, and FOBT/FIT in the same calendar year. The exclude veterans with evidence of prior colonoscopy within 10 years, of Disease (9th and 10th edition) diagnostic code or by self-report. We will also Exclusion criteria: Have any known gastrointestinal symptoms such as bleeding, unexplained weight loss, or change in bowel habits, family history of CRC, inflammatory bowel disease (IBD), or colectomy using International Classification
- ġ. List all screening and/or eligibility requirements.
- study but who have not been seen by primary care in the past 18 months prior to Men and women veterans age 50-75 on the date of screening for eligibility Received care in the CMCVAMC in the 18-48 months prior to selection for the
- Are due for screening
- ₹ are asymptomatic for CRC
- < prior 5 years, and FOBT/FIT in the same calendar year. Have no evidence of colonoscopy in the prior 10 years, sigmoidoscopy in the
- ≤. inflammatory bowel disease (IBD), or colectomy unexplained weight loss, or change in bowel habits, family history of CRC Have no history of any known gastrointestinal symptoms such as bleeding

or chart audits.) (The information used to exclude patients will be derived from the electronic queries

- ? colorectal cancer outside the VHA yet undocumented in VistA undergo a telephone interview to determine if they have received screening for before they are actually determined to be eligible for the study. Some patients may Explain any special test or evaluations potential subjects may have to undergo
- Not Applicable; subjects not recruited; chart review.
- ω If applicable, indicate what populations will be targeted for recruitment as participants. Check all that apply.

| Not Applicable, chart review | Other (Specify) | Non-Veterans*** | Veteran Family members*** | Non-English Speaking** | VA Employees | Outpatients | Inpatients | Females | Males |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | $\boxtimes$ | | $\boxtimes$ | $\boxtimes$ |

a. \*\*For non-English speaking subjects - If an investigator proposes to use a participant Translator certification is also required. as well as the English version, needs to be forwarded to the IRB for approval. population that does not speak or read English, a copy of the translated document,

| b. ***If non-veterans will be recruited for this study, explain why sufficient veterans are not available to participate in the project (IVHA Handbook 1200.5, paragraph 16a). Veteran's spouses/partners, caregivers, etc. are considered non-veterans for the purposes of this study. ***What is the project larget a specific race or ethnic group as participants?** I Not Applicable ii. Ponting (Mon-veteran forms should be used IRB office will obtain approval from ACOS/R&D and Medical Center Director.) Does this project target a specific race or ethnic group as participants? I If yes, check all that apply. Race I If yes, check all that apply. Children (Under 18) Requires Waiver from CRADO (VHA) Directive 2001-028. Research Involving Children) Voung Adultis (18-21) Author (18-21) Author (18-21) Author (18-21) Author (18-21) Author (18-21) Are there specific reasons why certain population flat is eligible for routine specify reasons. We are studying a population that is eligible for routine specify reasons. We are studying a population that is eligible for routine and the project require enrollment of the following classes of participants? Express and participants? Express a participants? Vers No. Children (Under 18) Requires who are younger than 50 years or older than 75 years will not be included in our study. Race Conomically and/or educationally disadvantaged persons I prisoners I fermicity I patients I frace or ethnic groups a participants? VES NO. Enployees Individuals with impalied decision making capability Prisoners I prisoners I prisoners I prisoners I prisoners I prisoners are prisoned to recurrent groups or older than 75 years or older who are because or older who are because or older than 50 years or older who are because or older who are beca |
|---|

- generally postmenopausal. Thus, it is unlikely for a pregnant to be included in the
- ġ. project-specific measures or special considerations, steps, or safeguards to ensure that these individuals are adequately protected. Not applicable. See above. If the project requires enrolling any of the above classes of participants describe any
- Ω plan to randomize 783 patients. criteria. There are an estimated 3,388 potentially eligible veterans for this pilot, and we support from Dr. Tzanis, for participation and to confirm the inclusion and exclusion PCP approval, through discussion at scheduled clinical and program meetings with and not currently up-to-date on CRC screening in the beginning of 2016. We will obtain received medical care at CMCVAMC in the 18-48 months prior to the start of our study To summarize, we will run the electronic query to identify age-eligible veterans who had Patient selection for the study will be based on the criteria described in above sections. Describe the exact plan how subjects will be identified and recruited for the study
- advertisements and brochures. We will obtain PCP approval, through discussion at scheduled clinical and program meetings with support from Dr. Tzanis, for participation and to confirm the inclusion and exclusion criteria. Discuss methods, e.g., referrals from physician offices, clinics, programs, or through
- Ö information will be transmitted to the research staff. Not applicable If using a clinic, be specific about who will identify the potential subject and how that
- ဂ be recruited. Not applicable If snowball method will be used, discuss the process and how the first individuals will
- d The information to be sent to subjects will be included as part of the outreach kit flyers and advertisements (include all recruitment materials with this submission). Describe how information will be disseminated to subjects, e.g. handouts, brochures,

### Informed Consent

- a. Informed Consent will not be sought.
- Ö We are submitting the Oral Informed Consent Form instead of Written Form10-1086. Written informed consent from participants (VA Form 10-1086 is attached). Note:
- ဂ as required by VA policy and/or applicable state laws (VA Form 10-1086 is attached) Written informed consent from participants' legally authorized representative (LAR)
- Q Request Waiver of Documentation of Informed Consent 🛛
- Φ List the title of the key personnel involved in the following activities
- Person Obtaining Consent
- (a) ) Research Assistants
- be trained in the study procedures and have appropriate VA appointment Type of training received to perform this process: Research Assistant will Subjects certification including required VA information security training and have Human
- =: criteria described above medical records to prescreen patients for eligibility for the study based on the determine populations and individuals eligible for the study). We will use the Pre-Recruitment Screening (the use of medical records and other data bases to
- ≣ introduced to the study and to the possibility of participating as subjects): Not Recruitment Process (the process in which individuals are contacted and first
- ₹. consent for participating), We waiver of informed consent above informed about participating in the study and then formally give their voluntary Informed Consent Process (the process by which recruited subjects are fully


- < on review of EMR/CPRS. other person-specific information), The final decision on eligibility will be based phases of the study, using laboratory data, inclusion and exclusion criteria, and determination of eligibility of prospective subjects is made during the early Screening of Recruited Subjects (those activities in the protocol in which a final
- ς. Include the breakdown of each individual's responsibilities:
- (a) Principal Investigator, Supervision
- ﻕ Co-Principal Investigator, Supervision and selection of sample
- obtaining oral informed consent, and conducting phone interviews (d) Additional research staff by title, Dataset Manager/Analyst will select a list of Research Assistants, Determining eligibility through CPRS audits and
- potentially eligible patients from CPRS
- Will informed consent be obtained from potential subjects prior to determining LYES ⊠ NO \_ N/A
- involves procedures that are used in routine clincal care informed consent on over 3,000 patients prior to determining eligibility. The study Disclosure of Protected Health Information. It will not be feasible to obtain If no, provide justification and a HIPAA Waiver of Individual Authorization for
- ġ. they are considered enrolled on the study. Define when a subject is enrolled into the study, e.g. after the subject signs the informed consent or after randomized to treatment. Once a subject is randomized,
- h. Describe:
- privacy. not applicable, waiver of informed consent obtained The process when informed consent will be obtained and protecting patients
- consent. not applicable, see above Any waiting period between informing the prospective participant and obtaining
- compensation is provided. Steps taken to minimize the possibility of coercion or undue influence. No
- . Provide the language
- i. Used by those obtaining consent not applicable
- **English or Spanish** Understood by the prospective participant or the legally authorized representative
- Provide location where informed consent will be obtained. not applicable
- 10. Waiver or Alteration of Informed Consent Requirements/Waiver of Requirement to **Obtain Documentation of Informed Consent** Are you requesting a waiver or alteration of informed consent? (Check all that apply)
- participate will likely represent those willing to return the kits. We will therefore research infeasible and alter the design because individuals who consent to waiver. In this pragmatic study, we are seeking to determine optimal approaches dedicated staff. Therefore, a waiver will not adversely affect the rights and practices of screening by informing patients by phone of test results with a to deliver colorectal cancer screening. Getting consent will inherently make the welfare of the subjects. The research cannot be practically carried out without the increasing the reach of screening to veterans. We will also enhance the current required outside of the research context. The study offers a net benefit in subjects and involves no procedures for which written consent is normally settings. Thus, the research presents no more than minimal risk of harm to care for delivering colorectal cancer screening in the VA and in a variety of other The procedures to be used involve methods that are currently the standard of Yes; provide justification. M This research involves no more than minimal risk.

011

of screening in the VA, compared to the current usual care. the study. For instance, all selected subjects will receive information about CRC screening including the testing options (see attached for examples). This pilot program is designed to effectiveness of mailed FIT outreach to increase the use invitation to screen. Subjects will receive additional pertinent information about screening will likely consent. This will undermine our ability to test the study. The bias occurs because only subjects interested in colorectal cancer hypotheses. We are interested in the proportion of individuals who respond to the the VA. This will lead to a serious selection bias and lead to a fatal flaw in the not be able to learn from those unwilling to participate in screening, a priority for

 b. Yes; for recruitment purposes only. Are you requesting a waiver to obtain documentation of informed consent? Yes; provide justification. ⊠ (a) An IRB may waive the requirement for the investigator to obtain a signed (e) (a)  $\boxtimes$  1. The research involves no more than minimal risk to the subjects; (b)  $\boxtimes$  2. The waiver or alteration will not adversely affect the rights and welfare documents that: waive the requirements to obtain informed consent provided the IRB finds and An IRB may approve a consent procedure which does not include, or which alters, some or all of the elements of informed consent set forth in this section, or <u>a</u> <u>බ</u>  $\equiv$  $\boxtimes$  3. The research could not practicably be carried out without the waiver or consent form for some or all subjects if it finds either:

(i) 1. That the only record linking the subject and 4. Whenever appropriate, the subjects will be provided with additional (iv) Possible changes in methods or levels of payment for benefits or services (iii) Possible changes in or alternatives to those programs or procedures; or evaluate, or otherwise examine: to the approval of state or local government officials and is designed to study, alteration; and of the subjects; pertinent information after participation 5. The research or demonstration project is to be conducted by or subject  $\boxtimes$  2. That the research presents no more than minimal risk of harm to Public benefit or service programs; NOTE: In cases in which the documentation requirement is waived, the subjects and involves no procedures for which written consent is normally whether the subject wants documentation linking the subject with the resulting from a breach of confidentiality. Each subject will be asked the consent document and the principal risk would be potential harm under those programs. Procedures for obtaining benefits or services under those programs; required outside of the research context. research, and the subject's wishes will govern; or written statement regarding the research IRB may require the investigator to 1. That the only record linking the subject and the research would be provide subjects with a

0

- S Compensation (The amount of compensation may not constitute an undue inducement to participate in the research.
- financial or other compensation provided for participation in the study Summarize any financial compensation that will be offered to subjects. There is no


- N Provide the schedule for compensation. No compensation is provided
- Per study visit or session. None
- Total amount for entire participation. None
- Explain how compensation will be provided via cash, voucher, gift card, etc. Not applicable
- 40 If financial compensation will be prorated, explain the process. Not applicable
- Not Applicable -

### $\exists$ Withdrawal/Early Withdrawal

- months after baseline can withdraw from participation by stopping the survey questions program. We will adopt this approach for the proposed program. Subjects contacted 6 usual approach is to place such subjects on a 'do not contact' list for the specific not uncommon in screening programs for some subjects to opt out of screening. The the pragmatic trial will be asked to contact the office to report their eligibility status. It is Describe how and when a subject may withdraw from the study. Those included in
- Ņ advised when called that they can withdraw from the study at any time. Provide procedures for the orderly termination of participation by the participant and if any consequences would result from early withdrawal from the study. There are no consequences associated with withdrawal from the study. Subjects will be
- ω Explain if survival data is required. If so, clarify how data will be obtained. Not
- 4 Not Applicable; subjects not recruited; chart review.

### $\subseteq$ Risk/Benefit Assessment

## **Potential Study Risks**

- Describe and assess all of the following risks that may be associated with the
- Physical There is no risk of physical harm to participants
- with primary care doctors to ensure that diagnostic work up is addressed by the results to ensure that diagnostic testing is performed and coordinate our efforts will also be trained to elicit any concerns the patient may have and encourage the patient to schedule the appointment. We will also track patients with positive with cancer. We are addressing this by training the Research Assistants to facilitate timely scheduling of diagnostic colonoscopy. The Research Assistants receiving a positive screening result. This may create anxiety about diagnosis primary care doctor. Psychological There is minimal risk of psychological harm resulting from
- ≣ Social There is minimal to no risk of social harm from this study
- ₹ may provide economic benefit from the averted cost and morbidity of late-stage cancer treatment. Economic There is minimal to no risk of economic harm. Early detection of CRC
- < *Monetary* None
- ≤ Legal None
- study materials are inadvertently disclosed or stolen. In discussing with the that our procedures are JCAHO-compliant. purposes of identifying the patient. We will explore this option, but also ensure CMCVAMC Lab Director, using an order number may be sufficient for the Loss of confidentiality. There is a small risk of loss of confidentiality if PHI or
- viii. Assess the likelihood and seriousness of such risks. This is addressed under each section above.

- Ö approved mailing methods. methods are routinely used in clinical settings including the VHA and we will use VA loss of confidentiality while the test is being mailed to patients. However, our that are consistent with each individual's job description. There is also the risk of Permissions of research staff on the project will be reviewed periodically to ensure and only trained authorized personnel will be allowed access to the patient data. identification numbers will be kept in a secure location in password-protected drives, procedure to mail kits to patients. The crosswalk file containing patient study following VA information security procedure for data safety. We will use VA earliest available timeslot. We will reduce the risk of loss of confidentiality by minimal risk of psychological distress by helping to schedule a colonoscopy in the Specify what steps will be taken to minimize these risks. We address the small and
- ဂ screening program to patients, the study itself will be conducted within the existing CMCVAMC CRC were considered and why they will not be used. Our methods represent minimal risk If methods of research create potential risks, describe other methods, if any, that
- a stored in secure password-protected drives with access granted to authorize staff. Identifiable data will not be allowed to be removed from the VA and only de-identified data will be stored in research files at CHERP, CMCVAMC Center Annex (3900) Woodland Drive) Suite 202, file room 235 Philadelphia, PA 19104. receive VA Privacy and Information Security Awareness training; all data will be privacy policy and all research staff will have appropriate VA appointment and be taken to minimize these risks. As outlined above, we will adhere strictly to VA If chart review, breach of confidentiality is always a concern. Specify what steps will

### Ņ **Potential Study Benefits**

- potential benefit from the project and the risks to participants are minimal. If the subject does not receive any direct benefit, then it must be stated here and in stage cancers if undetected, unlike current strategies. Thus, there is substantial less likely to have regular medical visits and thus may be at risk for developing laterindividuals than colonoscopy. Our proposed approach can reach individuals who are screen individuals in a way that is non-invasive and may appear less threatening to less likely to be screened. This study provides a simple and inexpensive way to cancers early, and hence decreases the risk of CRC death. This is particularly important for minority populations who are at higher risk for the disease but may be FIT, which is inexpensive and has high sensitivity and specificity for detecting Assess the potential benefits to be gained by the individual subject, as well as is potentially preventable through screening and the VA recommends the use of the benefits that may accrue to society in general as a result of the planned work. CRC
- ġ. the consent form. Early cancer detection will be highly beneficial to patients

#### ω **Alternate Procedures**

- ability to do so will not be restricted by the study. Subjects can receive screening for colorectal cancer outside this program. Subjects' Describe the alternatives available to the subject outside the research context
- Þ applicable If none, state that the alternative is not to take part in this research study at all. Not

| | | .< |
|---|---|---|
| with any study.) | III studies are required to have a DSMB. However, the IRB has the right to require a DSMB | V. Data and Safety Monitoring Board (DSMB) or Data Monitoring Committee (DMC) (All Phase |
| | , the IRB has the right to require a DSMB | Monitoring Committee (DMC) (All Phase |

| :- | |
|-----------------------------------------------------------|---|
| Will an ir | |
| an | l |
| Will an independent DSMB or DMC oversee the project? ☐YES | |
| DSMB | |
| ᄋ | |
| DMC | |
| 9 | |
| ersee | |
| ₽ | |
| project? | |
| YES | |
| □<br>NO | |
| X<br>N<br>A | |

HRPP Approval: 06/15/2011
R&D Approval: 07/05/2011
File: K: New IRB Forms

| | | a. |
|---|---|---|
| i. Name: | Center Representative and attach a copy of the charter. | If yes, please provide contact information |
| Phone Number: | y of the charter. | information for the DSMB or DMC or Coordinating |

N If a DSMB or DMC will not monitor this study, who will monitor this study? Check all that

E-mail:

| <ul> <li>a. Principal Investigator</li> <li>b. Sponsor</li> <li>c. VA Cooperative Studies Program</li> <li>d. Safety monitoring committee</li> </ul> | | | | | |
|---|---|---|---|---|---|
| Principal Investigator Sponsor VA Cooperative Studies P Safety monitoring commit | ٩ | ი | ġ. | a. | 3 |
| | ty monitoring commit | tudies P | Sponsor | rincipal Inves | <u> </u> |

- .≤ Data Monitoring (Monitoring plans describe how a monitor, independent of the study team, center phase III trials. Federally funded studies may require the use of an independent DSMB.)

  1. Describe the data monitoring plan. (All protocols must have a data monitoring plan applicable research regulations and CMCVAMC requirements. Such independent boards are usually reserved for high-risk phase I studies, or large, multi necessarily require the use of an independent Data and Safety Monitoring Board (DSMB). regularly inspects study records to ensure the study is adhering to the study protocol and Monitoring plans do not
- occurrence in accordance with IRB guidelines and VA rules. oversight will be provided through the IRB at the VA. Any adverse events, e.g. evidence authorized staff will be provided access via password to study databases. Additional conducting regular data checks to ensure the accuracy of the data collected. Only Research staff will also have appropriate VA appointments such as a WOC and be required to complete VA Privacy and Information Security Awareness training and for use of EMR in clinical and observational studies. Thus, procedures for protecting patient data have become enhanced. The PI will provide oversight for all data collection immediately reported to study investigators and to the IRB within 24 hours of its of severe psychological distress as a result of news of a positive test result, will be manager will regularly monitor the database. included in the IRB protocol before beginning study activities. The PI and a database maintaining and updating a tracking REDCap database of screen-eligible individuals the Collaborative Institutional Training Initiative (CITI) and will be responsible for and analysis procedures. Research staff will have human subject's certification through we will make every effort to ensure the safety of all data collected. There is precedence ascertain response rates, and assess the ability to reach patients. Because this is NOT a study that involves an investigational drug or device, there will be no DSMB. overall progress of the study, ascertain how many subjects are identified/recruited, study quarterly to evaluate adherence to policy and overall progress. We will review the with the co-Investigators will monitor the study's data. We will review the progress of the appropriate for the potential risks and the complexity of the study.) In addition, research staff will assist in The PI in collaboration
- Ġ sponsor. (Refer to the CMCVAMC IRB Standard Operating Procedure (SOP) Manual Describe how protocol deviations, adverse events, serious adverse events be undertaken. PI, and appropriate actions as directed by the IRB including additional staff training will protocol deviations will be reported to the IRB within 1 hour of it becoming known to the unanticipated or unexpected problems will be reported to the CMCVAMC IRB and breaches of confidentiality, unanticipated adverse device effect (UADE), and for reporting guidelines.) Any breach of confidentiality, unanticipated problems, or
- protections such as: Describe the management of information obtain that might be relevant to participant


- within 1 hour and if necessary, patients will be referred to the appropriate clinical problems such as psychological problems in a subject will be reported to the IRB Unanticipated problems involving risks to subjects or others: Any unanticipated
- =: be adopted for routine clinical practice. effective than with current usual practice, the procedures under study is likely to If however our results show that screening using the outreach approach is more recommended once every year. Thus, there will be no need for interim analysis. Interim results: This is a 1-year study. Screening for CRC using FIT is
- procedure, or to add or remove staff. to make such changes as increase the number of study subjects, add a new Protocol modifications: When needed, we will seek modification of the protocol

## ω If applicable, define the plan for subjects if research shows results such as:

- a result of our study. However, if it occurs, the research assistants will be trained as services at the CMCVAMC. part of our standard operating procedures to refer the patient for mental health Depression There is a minimal risk of subjects developing or reporting depression as
- Suicide There is minimal to no risk of suicide occurring as a result of the study.
- 0 Abuse There is minimal to no risk of abuse being detected during the course of this

### Statistical Analysis

- participants could be ineligible post-randomization, we will recruit about 783patients invitation-reminder vs. mailed-FIT. Accounting for the possibility that up to 20% of reminder, and 152 patients per arm will give a power of 80% for the screening sample size of 500 (250 per arm) will give 80% power for UC vs. screening invitationwith invitation- reminders, and 40% with mailed FIT. With those assumptions, a total power and sample size analysis, we assumed 15% screening rate in UC alone, 25% those assigned to mailed-FIT completed screening compared to 12% in UC. In our Include statistical power calculations and the assumptions made in making these for the pragmatic trial. calculations. Gupta et al. found that, among underserved patients in Dallas, 40% of
- σ approach will be 'intention-to-treat' analysis and additional analyses will be restricted sociodemographic measures with the outcome of FIT completion. The primary alpha of 0.05) to examine associations of patient characteristics and We will use both univariate and multivariable logistic regression analyses (2-sided when the program is fully implemented, and if larger sample sizes will be needed understand if there are patient groups that may need specific targeted outreach race, which is consistent with our own experience. This analysis will allow us to found that screening use differed by age and was lower among persons of black such as marital status and other factors such as sex. Our rationale is that a VA study vs. 65+ and race/ethnicity as predictors, controlling for socio-demographic covariates test using logistic regression. We will focus primarily on age categorized as 50-64 completion of mailed FIT (dependent variable) among recipients of the mailed FIT outcome. We will assess the association of age and race/ethnicity with the tests other than FIT to warrant examining "receipt of any CRC screening test" as an test types to assess whether there are large enough numbers of patients receiving All tests will be based on a 2-sided alpha of 0.05. We will examine the distribution of mailed-FIT and invitation-reminder are equal using an "intention-to-treat" approach. hypothesis that the completion rates between the mailed-FIT and UC and between plan, stopping rules and endpoints. We will use Chi-squared statistic to test the null Define plans for data and statistical analysis, including key elements of the statistical

HRPP Approval: <u>06/15/2011</u>
R&D Approval: <u>07/05/2011</u>
File: K: New IRB Forms

| patterns of testing and screening rates and screening outcomes in the VA. | potential variation in rates of screening across the VA, and relate those to the | calling participants. We will also generate a report of the screening practices and | addresses or were unreachable. We will seek to verify addresses of returned mail by | characterize the proportion of invitees whose mail was returned due to bad | address is needed to conduct outreach to patients. Thus, it is important to | completion rate of mailed kits, as well as seasonality effects. A valid participant | relation of other factors such as socioeconomic status and place of residence on | to those with valid addresses. In future studies, we will be able to investigate the |
|---|---|---|---|---|---|---|---|---|

- × Privacy and Confidentiality (Privacy refers to persons and to their interest in controlling the unauthorized disclosure or intelligible interception.) (Investigator should contact the Privacy access of others to themselves.) (Confidentiality refers to protecting information from Officer for additional details.)
- apply. Indicate the type of data that will be received by the Principal Investigator. Check all that
- participant. (Contact Privacy Officer for assistance. If data is coded, it is not ceil De-identified – Without any identifiers that could link the data to a specific
- Ö considered de-identified.)

  Identified – Linked to a specific participant by identifiers sufficient to identify participants. (See HIPAA and Common Rule Criteria for list of identifiers.)
- 9 coded is checked, specify: participants. (See <u>HIPAA</u> and <u>Common Rule</u> Criteria for list of identifiers.)

  Soded – Linked to a specific subject by a code rather than a direct identifier. If
- subjects will be kept by the analyst/programmer and the PI Explain who will maintain the link or code. The code for identifying study
- subject for purposes of obtaining data or cleaning data. other staff will be granted access only when needed to identify specific research Richardson, and the Dataset Manager/Analyst will have access to the code. All Describe who will have access to the link or code. Only the PI, Drs. Doubeni,
- ≣ identifiers. However, analytic data will be stripped of all identifiers. Each subject will be identified using an encrypted unique identification number. The code or crosswalk file will be stored by the PI and the Dataset Manager/Analyst in a secure password-protected location. Provide exact details for how the data is coded. The study data will contain
- Does the project require the use of existing Protected Health Information (PHI) from a database, medical records, or research records? XYES NO NO
- If yes,

3

- the screening database used by Dr. Abraham Dubb. Specify the source of the existing PHI Clinical records in CPRS. We will also use
- ≓ numbers, etc.) on the below table. Indicate the specific data elements/identifiers (e.g., name, address, phone
- Ö If the study uses an existing database/data warehouse,
- VistA/CPRS supplemented by a clinical screening REDCap database used by Provide a description of the database/data warehouse. The study will use
- =: Dr. Dubb to identify patients and their screening history

  Make clear who is responsible for maintaining it. The REDCap database will be maintained by the Dataset Manager/Analyst with guidance from the PI in consultation with Dr. Abraham Dubb
- ≣ Cite any relevant Standard Operating Procedures (SOP) for the database/data These are existing VA standard databases
- Provide a copy of the SOP. These are existing VA standard databases
- ω Will PHI be collected prior to obtaining informed consent? ⊠YES ON O


- Disclosure of Protected Health Information with this submission. If yes, complete and provide a HIPAA Waiver of Individual Authorization for
- 4 or indirectly. HIPAA Identifiers - Indicate the PHI that will be collected from project participants directly
- C digits of a zip code if, according to the current publicly available data from the Bureau Name

  Name

  All geographic subdivisions smaller than a State, including street address, city,

  All geographic subdivisions smaller than a State, including street address, city, county, precinct, zip code, and their equivalent geocodes, except for the initial three of the Census All elements of dates (except year) for dates directly related to an individual, and
- except that such ages and elements may be aggregated into a single category of all ages over 89 and all elements of dates (including year) indicative of such age,

| Elephone numbers |
|---|
| tes 🖂 |
| tes |
| tes |
| tes |
| ces |
| IXI Telephone numbers |
| Fax numbers |
| Modical record much au |
| Though show the same to the sa |
| Health plan beneficiary numbers |
| Account Numbers |
| Certificate/license numbers |
| Vehicle identifiers and serial numbers, including license plate numbers |
| Device identifiers and serial numbers |
| Web universal resource locators (URLS) |
| Internet protocol (IP) address numbers |
| Biometric identifiers including fingerprints voiceprints audio recordings |
| المام |
| Full-face photographic images and any comparable images |
| The state of the s |
| Any other unique identifying number, characteristic, or code |
| Personal and Family History |
| ] |
| ☐ HIV (testing or inte |
| Disconstic/Laboratory tooks |
| ][ |
| :<br>:<br>:[ |
| . Ciller Records: |

Ģ Will participants be contacted from existing PHI? ⊠YES ON O

<

Ľ.

× ≤

ففدة

0

? 3

7.0

subjects). Patient selection for the study will be based on the criteria described in same information as listed under section R.8 identification and recruitment of If yes, clearly explain how participants will be contacted (NOTE: this would be the clinical and program meetings with support from Dr. Tzanis, for participation and to beginning of 2016. We will obtain PCP approval, through discussion at scheduled prior to the start of our study and not currently up-to-date on CRC screening in the above sections. To summarize, we will run the electronic query to identify age-eligible veterans who had received medical care at CMCVAMC in the 18-48 months

HRPP Approval: <u>06/15/2011</u>
R&D Approval: <u>07/05/2011</u>
File: K: New IRB Forms

- eligible veterans for this pilot, and we plan to randomize 783 patients. confirm the inclusion and exclusion criteria. There are an estimated 3,388 potentially
- 9 Principal Investigator, Co-Investigator, Statistician, Dataset Manager/Analyst, Research Provide the titles of the exact individuals who will have access to the collected data.
- access to the data for purposes of collecting, analyzing, interpreting, and Explain why these individual will have access to this data. These individuals need disseminating the results
- :< Information Security (Contact the Information Security Officer for additional assistance regarding confidentiality (storage/security) of research data.
- volume, it is feasible for us to confirm eligibility through chart audits prior to mailing patients during Months 3-5 of the study in weekly waves of about 50 mailings; with this Provide the precise plan how data is to be collected or acquired (repeat the same invitations to study participants. block-randomized to UC, invitation-reminder, or mailed-FIT with guidance from Dr. Richardson to achieve the desired sample size. We will mail all study materials to information as listed under "Data Collection" section of this form. Patients will be
- Participants randomized to UC: These patients will continue to receive the current participants in the trial, including those in UC, will receive follow-up of test results and will be embedded within this existing program for a pragmatic approach. However, all practice at CMCVAMC of offering screening during an office visit. Other interventions navigation to diagnostic colonoscopy for positive FIT results.
- σ week the invitation letter was sent (time zero). It is generally unclear whether mail colonoscopy, if needed. For the purposes of this intervention, Week 1 will be the invitation letter. They will also receive notification of test results and navigation to scheduled). They will receive three weekly reminders at weeks 4, 5, and 6 from the as change in bowel habit with rectal bleeding. The packet will also have a screening offered at CMCVAMC), and symptoms that should prompt diagnostic work-up such see below). The information will include lay-audience description of screening tests such as FIT and colonoscopy and, if appropriate, Cologuard (sigmoidoscopy is not information about CRC testing in the mail-FIT arm (except the kit and instructions, continue to receive UC. They will in addition receive an invitation letter with all of the Participants randomized to screening invitation-reminder: These patients will success of each approach used during the study. mailed reminders when participants cannot be reached by phone and track the may also change or a veteran may be homeless. Thus, we will also explore sending telephone numbers may change or run out of purchased minutes, but addresses reminders may be more effective at reaching veterans than phone calls because invitation letter if screening is not completed (even if they have an appointment letter will inform patients that a telephone reminder will follow in 4 weeks from believes he/she is not eligible and to update the contact information on record. The confirmation card and have instructions to contact the study team if the patient
- c with the invitation-reminder arm), followed by 2 additional calls at the end of weeks 5 receive a live telephone reminder (even if they have an appointment scheduled, as return their kit after 4 weeks of the date the pre-notification letter was mailed will weeks from notification letter if screening is not completed. Patients who do not information on record. They will be informed that a telephone reminder will follow 4 team if the patient believes he/she is not eligible and to update the contact week later (see section D2d2). Patients will receive instructions to contact the study (plus a screening invitation and screening confirmation card) followed by the kit 1 Participants randomized to Mailed-FIT will receive a mailed FIT pre-notification letter


HRPP Approval: 06/15/2011
R&D Approval: 07/05/2011
File: K: New IRB Forms

- approaches for successfully contacting participants in our study setting. the pre-notification letter was sent (time zero). We will explore and evaluate the and 6, if needed.82 For the purposes of this intervention, Week 1 will be the week
- a under the supervision of the PI in collaboration with Dr. Doubeni. Unless otherwise specified, data collection will be performed by a research assistant
- Φ. the PI and Drs. Richardson and Doubeni. The Dataset Manager/Analyst will perform analysis on the study with guidance from
- CHERP The research data obtained will be stripped of all identifiers prior to analysis at the
- N report forms, etc. limited to signed, original informed consent and HIPAA authorization forms, case Provide a listing of the exact research data that will be stored, including but not

The data to be collected are listed below in the table

| Measures | Definition and elements |
|---|---|
| Socio-demographics | Age, sex, race/ethnicity, education/SES/geocode, marital status |
| Contact information | Address, phone, next of kin, emergency contact, whether address is |
| | invalid |
| Access/Healthcare | PCP (name/type), usual place of care, visit history, transportation |
| utilization | |
| Eligibility for outreach | Eligible (Y/N), ineligibility reason and duration (permanently |
| | ineligible due to age, colectomy, IBD, CRC history, etc., or year |
| | when becomes eligible again |
| Risk factors/symptoms | Height/weight, family history, etc., GI symptoms |
| Screening history | Prior colonoscopy/sigmoidoscopy/FOBT/barium enema date and |
| | reason |
| Mailed introductory letter | Notified to expect the kit/general information about screening and |
| | CRC symptoms |
| Mailed kit | Dates FIT was mailed, date received |
| Reminders | Dates of reminders to return kit with a flag for those ineligible |
| Refusals | Date and reasons for refusal |
| Test collection | Date sample was collected by patient |
| Date test received and | Date kit was received and date tested (goal is within 72 hours) |
| tested | |
| Received some other | Received colonoscopy or other test instead of returning FIT, and |
| screening | results |
| FIT result/notification | Result (positive, negative, or incomplete), patient and provider |
| | notification dates and methods (mail, phone, electronic), and entry |
| | into EMR |
| Diagnostic testing | Receipt of colonoscopy for positive FIT, and results |
| Detected lesions | Number and types of lesions detected |
| Ambient temperatures | Ambient temperature on collection and receipt date from NOAA |
| | databases |
| Cancer registry (linkage | Date, stage, morphology, behavior, grade, & location |
| only) | |

ω team members. A master copy will be stored and copies created for analytical purposes protected and will be only accessible to the PI, analysts and other authorized research provide corresponding security systems. All data will be stored in secure network Indicate how project's research data (original and all copies) will be stored and


HRPP Approval: <u>06/15/2011</u>
R&D Approval: <u>07/05/2011</u>
File: K: New IRB Forms

will be conducted in accordance with VA privacy policies Room 235, 3900 Woodland Drive, Philadelphia, PA 19104 All data storage procedures Paper copies will be stored at the CMCVAMC CHERP: Center Annex Suite 202, File

- 4 Health Equity Research and Promotion (CHERP), Center Annex (3900 Woodland Computing Infrastructure [VINCI] server workspace under the auspices of the Center for CMCVAMV. De-identified research data will be stored in the VA Informatics and will be stored and secured. Identifiable data will remain behind firewalls at the CMCVAMC, provide exact location where research data (original and all copies) Avenue Philadelphia, PA 19104) Suite 202 Cubicle #9.
- Ç Data will not be transmitted, but rather stored in network drives that are accessible from Explain how data is to be transported or transmitted from one location to another. within the VA, both at the main campus and at CHERP at the Philadelphia VA Medical

| <ul> <li>a. Informed Consent discloses PHI transported or transmitted off-site. ☐YES ⊠NO ☐N/A</li> <li>b. HIPAA Authorization discloses entities to which PHI will be transported or</li> </ul> | ဂ္ဂ န | Within the va, both at the main campus and at offern at the rimadelphia va wedicar<br>Center Annex |
|---|---|---|
| □N/A HIPAA Authorization discloses entities to which PHI will be tran | • | Informed Consent discloses PHI transported or transmitted off-sit |
| <ul> <li>HIPAA Authorization discloses entities to which PHI will be tran</li> </ul> | | □N/A |
| | | HIPAA Authorization discloses entities to which PHI will be trans |

0.0 If yes, list the exact data that will be transmitted. Not applicable

and the justification for such disclosure and the authority.

List all entities or individuals outside CMCVAMC to whom data is to be disclosed,

- If yes, explain how data will be protected during transmission outside of CMCVAMC
- Φ Off-site, provide exact location Not applicable (If off-site, attach at least one of the

| ≓ | ≓ | | 0 |
|---|---|---|---|
| Memorandum of Understanding ☐YES ☐NO ☒N/A | Off-Site Storage/Transfer of Research Data ☐YES ☐NO | Data Use/Transfer Agreement ☐YES ☐NO ☒N/A | ĺ |
| | N/A | | |

- ₹ (Note: VA data disclosed to a non-VA investigator at an academic affiliate for research purposes needs to be approved by the Under Secretary of Health or designee.)
- 6 List who is to have access to the data and how they are to access it (anyone who has access to the data is responsible for its security).
- Doubeni, Chyke
- Richardson, Diane M.
- 9 Dataset Manager/Analyst
- Research Assistants
- 7 **information** (e.g., the Coordinating Center, the statistician, and PI who has ultimate responsibility). The PI, dataset manager/analyst, statistician (Diane M. Richardson), Dr. Describe who is to have access and be responsible for the security of the
- 00 on the shared folder. Regular reviews will be conducted to ensure that appropriate manager/analyst will control who has access to the data. They will assign permissions Provide mechanisms used to account for the information. The PI and dataset permissions remain in place.
- 9 Give security measures that must be in place to protect individually identifiable these policies. Identifiable information will be used only for the approved purposes privacy policies. We will seek guidance from the privacy officer when needed to develop information if collected or used. The use of identifiable information will follow VA

HRPP Approval: 06/15/2011
R&D Approval: 07/05/2011
File: K: New IRB Forms

- 10. How and to whom a suspected or confirmed loss of VA information is to be reported. Any suspected or confirmed loss of information will be reported by phone and letter to the IRR chair and VA privacy officer within 1 hour.

| 19. | 18. | | 16.<br>17. | 15. 14. | <del>1</del> 3. | | | 75 | <b>≓</b> |
|---|---|---|---|---|---|---|---|---|---|
| one hour of the improper use or disclosure. 19. <b>Is there a plan to apply for a Certificate of Confidentiality?</b> ☐YES ☒NO ☐N/A a. If yes, provide a copy of the certificate with this application or to the IRB Office as | Descri<br>All rese<br>user-lev<br>a. The | <ul> <li>(FISMA) standards.</li> <li>a. Data is stored: <ol> <li>i. With identifiers - □YES ☒NO</li> <li>ii. Coded - ☒YES □NO</li> <li>iii. De-Identified - ☒YES □NO</li> <li>iv. Provide the exact list of identifiers that will be stored. Encrypted study</li> </ol> </li> </ul> | | | | <ul> <li>added to an amended protocol for IRB review prior to the start of research.</li> <li>ii. External drive that is password protected and/or encrypted. □YES ⊠NO □ N/A</li> <li>(a) If yes, identify the external drive.</li> <li>c. Off-Site server □YES ⊠NO □N/A (If off-site, attach at least one of the following.)</li> </ul> | - O - A | and describe appropriate actions to provide such safeguards. This study does not involve vulnerable populations. All subjects will receive the same information and/intervention based on the study arm each subject is assigned to. Electronic PHI will be stored on the following: | rights and welfare of subjects who are likely to be vulnerable including, but not |

HRPP Approval: <u>06/15/2011</u>
R&D Approval: <u>07/05/2011</u>
File: K: New IRB Forms

soon as received.

### 20. Record Retention:

- until disposition instructions are approved by the National Archives and Records VHA Handbook 1200.05 §26.h Administration and are published in VHA's Records Control Schedule (RCS 10-1). The required records, including the investigator's research records, must be retained
- Þ Until a schedule for local research records is published, ALL records including Modifications Addressing VA Record Retention Requirements (July 23, 2009) identifiers must be retained." ORO/ORD Guidance on Informed Consent Form
- S If there are additional procedures for record retention, explain further.

## Qualification of the Investigators:

- Provide a description of the qualifications of each Investigator/Co-Investigator and their specific role in the study.
- processes of care and outcomes on CRC, including at the VA. colorectal surgery. She is a clinical epidemiologist whose research focuses on member of the Department of General Surgery at CMCVAMC with clinical practice in in the Perelman School of Medicine at the University of Pennsylvania (UPenn) and a E. Carter Paulson, MD, MSCE is the PI of the project. She is an Assistant Professor
- Þ at Kaiser Permanente. His research focuses on health disparities, the effectiveness multiple PI and chair of the CRC working group of the PROSPR (Prospective Research Optimizing Screening through Personalized Regimens) Research Center Medicine at Upenn, full member of the Abramson Cancer Center at Penn, and is general preventive medicine/public health and family medicine, is Chair of the Chyke A. Doubeni, MD, FRCS, MPH (Co-Investigator) is board-certified in both Department of Family Medicine and Community Health in the Perelman School of
- 9 investigator for several studies evaluating healthcare quality and disparities in outcomes. She has expertise in analyses of longitudinal and multilevel data, and design and analysis of RCTs. effectiveness study of influenza vaccination, and a statistical collaborator and Co-Biostatistics and Informatics Core, Core Investigator and Lead Biostatistician at the of screening, and improving the screening process for CRC. Diane M. Richardson, PhD (Co-Investigator/Statistician) is Co-Chief of the VA Center for Health Equity Research and Promotion, PI for a VA comparative
- Ņ If applicable, the Principal Investigator must identify a qualified clinician to be responsible for all study related healthcare decisions. Drs. George Tzanis and
- ω PI should submit a current, dated CV with each new initial review